CLINICAL TRIAL: NCT04835636
Title: A Pilot of a Modified Diabetes Prevention Program in Quito, Ecuador
Brief Title: Modified Diabetes Prevention Program in Ecuador
Status: Completed | Type: Observational
Sponsor: Ohio University (Other)
Collaborators: Touro University, California (Other)
Responsible Party: Sponsor
Other Study IDs: OHTU2021
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Diabetes Prevention Program — This program is a 1 year lifestyle modification program focused on reducing calories and fat calories and increasing physical activity to achieve a 7% weight loss. This study utilized the first 16 sessions (6 months) of the program

SUMMARY:
This pilot study will evaluate the use of a modified (cultural and language) adaptation of the National Diabetes Prevention Program in a cohort in Quito Ecuador.

DETAILED DESCRIPTION:
This pilot study will evaluate the use of a modified (cultural and language) adaptation of the National Diabetes Prevention Program in a cohort in Quito Ecuador. People who took the program had the option to participate in the research component. All participants selected the research component.

Adaptations- the coaches will be physicians from PUCE and they will administer this program for eligible employees who have biochemical prediabetes.

The program will be modified to be able to fit within the school curriculum. The diabetes prevention program will be offered in Spanish and the content modified to better fit the cultural norms for the Quito Ecuador population.

Participants will be adults with prediabetes as screened by the CDC Diabetes Risk Test and confirmed by HbA1c.

Outcome measures will include change in mean HbA1c, change in weight, physical activity, and attendance to the program.

ELIGIBILITY:
Inclusion Criteria: Adults who worked at the university and had biochemical prediabetes.

-

Exclusion Criteria: Those with known diabetes, those unwilling to complete a 6 month intervention.

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The faculty and staff at PUCE University in Quito Ecuador were invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
HbA1c | 90-120 days
  measure of glucose over 90-120 days

SECONDARY OUTCOMES:
Weight change | 6 months
  change in weight over the 6 month program

CONTACTS AND LOCATIONS:
Overall Officials: Jay H Shubrook, DO, Study Director — Ohio University/Touro University California

IPD SHARING:
Plan to Share IPD: No
We will not share any patient identifier information with anyone outside the study.